CLINICAL TRIAL: NCT00554710
Title: The Ideal Management of Crohn's Disease: Top Down Versus Step Up Strategies. A Prospective Controlled Trial in the Benelux
Brief Title: Top Down Versus Step Up Strategies in Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other)
Collaborators: Centocor BV (Industry); Schering-Plough (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P01872
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2007-11

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; immunomodulators; biologicals
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Azathioprine; Methylprednisolone; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients received three infusions of infliximab 5 milligrams per kilogram (weeks 0, 2 and 6) in combination with azathioprine 2-2.5 milligrams per kilogram per day from day 0 onwards. If the patients responded and tolerated both drugs, azathioprine was continued for the duration of the trial. Patients who were intolerant to azathioprine received methotrexate at an initial dose of 25 milligrams administered subcutaneously each week for 12 weeks with dose reduction to 15 milligrams per week thereafter. Following initial therapy, patients who developed worsening symptoms were retreated with additional infusions of infliximab. If symptoms persisted methylprednisolone was initiated and azathioprine or methotrexate was continued.
  Interventions: Drug: infliximab+azathioprine
- 2 (Active Comparator): Induction with methylprednisolone (MP) or budesonide (BUD): MP 32 mg/day for 3 weeks was followed by tapering by 4 mg per week to 0; BUD 9 mg per day for 8 weeks with tapering to 0 by 3 mg per week thereafter.Patients who worsened during the tapering had the dose increased to the initial dose and tapered again. If patients worsened, azathioprine (2-2.5 mg per day) was introduced. Patients who relapsed following withdrawal of steroids received a second course in combination with azathioprine. For patients who failed 4 weeks of steroids, MP dose was given at 64 mg/day for 2 weeks, tapered by 8 mg per week; azathioprine was added. Patients who remained symptomatic despite 16 weeks of azathioprine received infliximab (5 mg/kg IV at weeks 0, 2 and 6). Patients who relapsed despite methotrexate or those intolerant to both azathioprine and methotrexate also received infliximab, without antimetabolite therapy. Infliximab was repeated upon relapse of symptoms in these patients.
  Interventions: Drug: methylprednisolone or budesonide

INTERVENTIONS:
Drug: infliximab+azathioprine — infliximab 5 mg/kg at week 0,2 and 6 + azathioprine 2-2.5 mg/kg
  Other Names: remicade/imuran
  Arms: 1
Drug: methylprednisolone or budesonide — methylprednisolone 32 mg followed by taper or budesonide 9 mg/day followed by taper
  Other Names: Medrol, entocort, budenofalk
  Arms: 2

SUMMARY:
The study prospectively compares two treatment algorithms for newly diagnosed Crohn's disease: one 'aggressive' treatment with early introduction of immunomodulators and biologicals and one 'standard treatment' with corticosteroids and only later introduction of immunosuppressives and biologicals if disease activity requires that.

DETAILED DESCRIPTION:
This two year open-label randomized trial compares the early use of combined immunosuppression to conventional management in patients with active Crohn's disease who have not previously received glucocorticoids, antimetabolites, or infliximab. Patients assigned to combined immunosuppression receive azathioprine and 3 infusions of 5 milligrams per kilogram of body weight of infliximab at weeks 0, 2, and 6. Retreatment with infliximab and, if ultimately necessary, corticosteroids are used to control disease activity. Patients assigned to conventional management receive corticosteroids followed, in sequence, by azathioprine and infliximab. The primary outcome measure is remission without corticosteroids and without bowel resection at weeks 26 and 52.

ELIGIBILITY:
Inclusion Criteria:

* age 16 - 75 years
* diagnosis of Crohn's disease within the past 4 years
* no previous treatment with corticosteroids, antimetabolites, or biologic agents.
* Active Crohn's disease, defined by a Crohn's Disease Activity Index (CDAI)20 score of greater than 200 points for a minimum of 2 weeks prior to randomization.

Exclusion Criteria:

* immediate need for surgery
* symptomatic stenosis or ileal/colonic strictures with prestenotic dilatation;
* signs, symptoms or laboratory tests indicating severe, medical disease;
* documented chronic infection
* a positive stool culture for pathogens
* a positive tuberculin test or a chest radiograph consistent with tuberculosis.
* malignancy
* allergy to murine proteins
* pregnancy
* substance abuse

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2001-05; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
remission without corticosteroids and without surgical resection | month 6 and 12 after inclusion

SECONDARY OUTCOMES:
the time to relapse after successful induction therapy | within 24 months
the proportion of patients receiving infliximab, methylprednisolone and antimetabolites | within 24 months
the median serum C-reactive protein concentration | 24 months
the proportion of patients experiencing adverse events | 24 months
the mean endoscopic severity scores and the proportion of patients without ulcers | after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Geert R DHaens, MD, PhD, Principal Investigator — Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW
Locations (1):
- Imelda GI Clinical Research Center, Bonheiden, Belgium

REFERENCES:
- [Derived] D'Haens G, Baert F, van Assche G, Caenepeel P, Vergauwe P, Tuynman H, De Vos M, van Deventer S, Stitt L, Donner A, Vermeire S, Van De Mierop FJ, Coche JR, van der Woude J, Ochsenkuhn T, van Bodegraven AA, Van Hootegem PP, Lambrecht GL, Mana F, Rutgeerts P, Feagan BG, Hommes D; Belgian Inflammatory Bowel Disease Research Group; North-Holland Gut Club. Early combined immunosuppression or conventional management in patients with newly diagnosed Crohn's disease: an open randomised trial. Lancet. 2008 Feb 23;371(9613):660-667. doi: 10.1016/S0140-6736(08)60304-9. PMID 18295023